CLINICAL TRIAL: NCT05457205
Title: Transcutaneous Spinal Stimulation for Reducing Lower Limb Spasticity in Chronic Spinal Cord Injury: a Cross-over Study of Immediate Effects and Outcomes of Home-based Therapy Trials
Brief Title: Transcutaneous Spinal Stimulation for Lower Limb Spasticity in Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Methodist Rehabilitation Center (Other)
Responsible Party: Principal Investigator, Matthias J. Krenn, PhD, Assistant Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UMMC-IRB-2022-9
Record Dates: First submitted 2022-07-05; First posted 2022-07-13 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries; Spasticity, Muscle
Keywords: Transcutaneous Spinal Cord Stimulation; Neuromodulation; Electrical Stimulation; Spasticity; Lower Extremities
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Neuromodulation with 50 Hz and low intensity (Experimental): Transcutaneous spinal stimulation for 30 min with a stimulation frequency of 50 Hz and stimulation intensity of 0.45 x lowest motor threshold (reflex threshold in leg muscles).
  Interventions: Other: Electrical neuromodulation
- Neuromodulation with 50 Hz and high intensity (Experimental): Transcutaneous spinal stimulation for 30 min with a stimulation frequency of 50 Hz and stimulation intensity of 0.90 x lowest motor threshold (reflex threshold in leg muscles).
  Interventions: Other: Electrical neuromodulation
- Neuromodulation with 100 Hz and low intensity (Experimental): Transcutaneous spinal stimulation for 30 min with a stimulation frequency of 100 Hz and stimulation intensity of 0.45 x lowest motor threshold (reflex threshold in leg muscles).
  Interventions: Other: Electrical neuromodulation
- Neuromodulation with 100 Hz and high intensity (Experimental): Transcutaneous spinal stimulation for 30 min with a stimulation frequency of 100 Hz and stimulation intensity of 0.90 x lowest motor threshold (reflex threshold in leg muscles).
  Interventions: Other: Electrical neuromodulation

INTERVENTIONS:
Other: Electrical neuromodulation — Electrical neuromodulation intervention using transcutaneous spinal stimulation: two self-adhesive semicircle electrodes (forming a 5cm round electrode) will be centered midline over the T11-12 spinal processes, and two 8×13 cm electrodes will be placed paraumbilical and interconnected to serve as a counter electrode. A current-controlled stimulator will deliver symmetric biphasic pulses (500-μs/phase). Electrical stimulation will be applied according to the description in each study arm.
  Other Names: Transcutaneous spinal stimulation; Transcutaneous spinal cord stimulation

SUMMARY:
Spasticity develops months after spinal cord injury (SCI) and persists over time. It presents as a mixture of tonic features, namely increased muscle tone (hypertonia) and phasic features, such as hyperactive reflexes (hyperreflexia), clonus, and involuntary muscle contractions (spasms). Spasticity is often disabling because it interferes with hygiene, transfers, and locomotion and can disturb sleep and cause pain. For these reasons, most individuals seek treatments for spasticity after SCI. New developments in electrical neuromodulation with transcutaneous spinal stimulation (TSS) show promising results in managing spasticity non-pharmacologically. The underlying principle of TSS interventions is that the afferent input generated by posterior root stimulation modifies the excitability of the lumbosacral network to suppress pathophysiologic spinal motor output contributing to distinctive features of spasticity. However, the previous TSS studies used almost identical protocols in terms of stimulation frequency and intensity despite the great flexibility offered by this treatment strategy and the favorable results with the epidural stimulation at higher frequencies. Therefore, the proposed study takes a new direction to systematically investigate the standalone and comparative efficacy of four TSS interventions, including those used in previous studies.

Our central hypothesis is that electrical neuromodulation with the selected TSS protocols (frequency: 50/100 Hz; intensity: 0.45 or 0.9 times the sub-motor threshold) can reduce and distinctly modify tonic and phasic components of spasticity on short- and long-term basis. We will test our hypothesis using a prospective, experimental, cross-over, assessor-masked study design in 12 individuals with chronic SCI (more than 1-year post-injury).

Aim 1. Determine the time course of changes and immediate after-effects of each TSS protocol on tonic and phasic spasticity. The results will reveal the evolution of changes in spasticity during 30-min of TSS and the most effective protocol for producing immediate aftereffects.

Aim 2. Determine the effect of TSS on spasticity after a trial of home-based therapy with each protocol. The participants will administer 30 min of TSS daily for six days with each of the four TSS protocols selected randomly. This aim will reveal the long-term carry-over effects of TSS intervention on various components of spasticity after SCI.

Aim 3. Determine the participants' experience with TSS as a home-based therapy through focus group meetings. We will conduct focus group meetings after participants finish the home-based therapy trial. Accomplishing this specific aim will provide a valuable perspective on the value, challenges, and acceptability of TSS as a home-based intervention.

The study addresses important questions for advancing scientific knowledge and clinical management of spasticity after SCI. Specifically, it will examine the efficacy of TSS frequencies and intensities on tonic and phasic spasticity. The study results will be relevant for a high proportion of individuals living with SCI that could benefit from this novel and low-cost non-pharmacological approach to managing spasticity after SCI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* History of SCI (ASIA Impairment Scale grades A-D)
* Time since injury longer than 6 months
* The presence of at least mild spasticity (>3) in the lower limbs by self-report of the Numerical Rating Scale (from 0 to 10) of spasticity severity
* Signed consent form

Exclusion Criteria:

* Neurological level of SCI below T11
* Suspected progression of SCI (e.g., syringomyelia)
* Ventilatory-dependent
* Implanted active devices (e.g., intrathecal baclofen pumps)
* Passive implants (plates, screws) between T10 and L3 vertebras
* Skin conditions precluding placement of electrodes
* Ongoing infections
* Pregnancy
* Difficulty following instructions
* No access to a caregiver/family member to help with electrode placement at home
* Other medical risks/contraindications as determined by the study physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-05 (Estimated)

PRIMARY OUTCOMES:
Change in posterior root reflex amplitude | Before and after an intervention session (30 minutes)
  The amplitudes of the posterior root reflexes will be calculated and normalized to the maximum response amplitude from the recruitment curve for each muscle separately. The respective values will be averaged over all muscles and used as an outcome measure.
Change in posterior root reflex amplitude (during intervention) | Before and during an intervention session (15 minutes)
  The amplitudes of the posterior root reflexes will be calculated and normalized to the maximum response amplitude from the recruitment curve for each muscle separately. The respective values will be averaged over all muscles and used as an outcome measure.
Change in flexion withdrawal reflex root-mean-square | Before and after an intervention session (30 minutes)
  The cumulative root-mean-square values of the reflex amplitude in a window from 50 to 200 ms after the stimulation pulse over all recorded muscles.
Change in flexion withdrawal reflex root-mean-square (during intervention) | Before and during an intervention session (15 minutes)
  The cumulative root-mean-square values of the reflex amplitude in a window from 50 to 200 ms after the stimulation pulse over all recorded muscles.
Change in pendulum test index | Before and after an intervention session (30 minutes)
  The pendulum test provides the spasticity index which is calculated based on the knee angle of the initial horizontal leg position of the pendulum test, the angle at which the leg reversed for the first time from flexion to extension, and the final knee resting angle.
Change in pendulum test index (during intervention) | Before and during an intervention session (15 minutes)
  The pendulum test provides the spasticity index which is calculated based on the knee angle of the initial horizontal leg position of the pendulum test, the angle at which the leg reversed for the first time from flexion to extension, and the final knee resting angle.

SECONDARY OUTCOMES:
Change in Modified Ashworth Scale | Before and after an intervention session (30 minutes)
  The total score will be obtained by summing the individual muscle scores (value 1.5 will be used for the 1+ scoring category). The sum score ranges from 0 to 40 (0, no increase in muscle tone across all 10 tested muscles).
Change in Modified Ashworth Scale (after one week) | Before and after one week
  The total score will be obtained by summing the individual muscle scores (value 1.5 will be used for the 1+ scoring category). The sum score ranges from 0 to 40 (0, no increase in muscle tone across all 10 tested muscles).
Change in Spinal Cord Assessment Tool for Spastic Reflexes | Before and after an intervention session (30 minutes)
  Sum of the 4-point scale of three types of spastic behavior (ankle clonus, flexor, extensor leg spasms).
Change in Spinal Cord Assessment Tool for Spastic Reflexes (after one week) | Before and after one week
  Sum of the 4-point scale of three types of spastic behavior (ankle clonus, flexor, extensor leg spasms).
Change in Penn Spasm Frequency Scale | Before and after an intervention session (30 minutes)
  Sum of spasm frequency (0-5 scale) and spasm severity (0-3 scale).
Change in Penn Spasm Frequency Scale (after one week) | Before and after one week
  Sum of spasm frequency (0-5 scale) and spasm severity (0-3 scale).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias J Krenn, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (2):
- United States (2):
  - Methodist Rehabilitation Center, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project information - Methodist Rehabilitation Center — https://www.researchmrc.org/projects/spinal-cord-injury